CLINICAL TRIAL: NCT02693678
Title: Real or Sham Diathermy vs Hand Massage in Lower Limbs Delayed Onset Muscle Soreness (DOMS) in Skiers, Effect on Knee Joint Proprioception
Brief Title: Real and Sham Diathermy vs Hand Massage in Lower Limbs Delayed Onset Muscle Soreness (DOMS)Effect on Knee Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Studi Fisioterapici di Montagna (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Lorenzo Visconti, PT, Studi Fisioterapici di Montagna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Studi FM
Record Dates: First submitted 2016-02-15; First posted 2016-02-29 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Musculoskeletal Pain
Keywords: Proprioception; Doms; Pain; Massage; Diathermy
MeSH Terms: conditions — Musculoskeletal Pain; Pain; Fever | interventions — Massage; Diathermy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Massage (Experimental): 10 min massage therapy with neutral cream on lower limbs following the patients indications, the points need to be related to the presence of DOMS
  Interventions: Other: Massage
- Diathermy (Experimental): 10 min diathermy with neutral cream on lower limbs following the patients indications, the points need to be related to the presence of DOMS
  Interventions: Device: DIathermy
- Sham diathermy (Sham Comparator): 10 min sham diathermy with neutral cream on lower limbs following the patients indications, the points need to be related to the presence of DOMS
  Interventions: Device: Sham diathermy

INTERVENTIONS:
Other: Massage
  Arms: Massage
Device: DIathermy
  Arms: Diathermy
Device: Sham diathermy
  Arms: Sham diathermy

SUMMARY:
Delayed onset muscle soreness (DOMS) can have an impact on the proprioception of knee joint . The study aim is to assess the effect of manual massage, diathermy and sham diathermy the proprioception of the knee joint in patients affected by DOMS.

DETAILED DESCRIPTION:
Delayed onset muscle soreness (DOMS) can have an impact on the proprioception of knee joint. The study aim is to assess the effect of manual massage, diathermy and sham diathermy on the proprioception of the knee joint in patients affected by DOMS.

Proprioception will be measured with "Technique" an App available on appstore , on the basis of the work on knee proprioception by S M Mir 2008 , and data about pain with numbering pain rating scale (NPRS) and pre-post treatment and global impression of change (PGIC) will be acquired.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DOMS after a skimountaineering race

Exclusion Criteria:

* Comorbidities, trauma

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Knee joint proprioception | 30min post treatment
  A video analysis of knee motion during a proprioception test will be done

SECONDARY OUTCOMES:
Patient global impression of change (partecipants can determine if after receiving the treatment they feel to be improved or not on an nominal level) | 30min post treatment
  A questionnaire will be submitted

OTHER OUTCOMES:
Numeric pain rating scale (NPRS) (1 to 10 scale where 1 is the minor level of pain and 10 is the worst) | 30min post treatment
  NPRS will be used

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Visconti, Principal Investigator — Studi Fisioterapici di Montagna

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mir SM, Hadian MR, Talebian S, Nasseri N. Functional assessment of knee joint position sense following anterior cruciate ligament reconstruction. Br J Sports Med. 2008 Apr;42(4):300-3. doi: 10.1136/bjsm.2007.044875. PMID 18390774
- [Background] Visconti L, Capra G, Carta G, Forni C, Janin D. Effect of massage on DOMS in ultramarathon runners: A pilot study. J Bodyw Mov Ther. 2015 Jul;19(3):458-63. doi: 10.1016/j.jbmt.2014.11.008. Epub 2014 Nov 24. PMID 26118518
- [Derived] Visconti L, Forni C, Coser R, Trucco M, Magnano E, Capra G. Comparison of the effectiveness of manual massage, long-wave diathermy, and sham long-wave diathermy for the management of delayed-onset muscle soreness: a randomized controlled trial. Arch Physiother. 2020 Jan 15;10:1. doi: 10.1186/s40945-019-0073-4. eCollection 2020. PMID 31956433